CLINICAL TRIAL: NCT05950048
Title: THE EFFECT OF WEB-BASED BREASTFEEDING COUNSELING GIVEN TO MOTHERS ON FULL BREASTFEEDING AND BREASTFEEDING MOTIVATION AND PROBLEMS
Brief Title: THE EFFECT OF WEB-BASED BREASTFEEDING COUNSELING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ayşe Gül KOCA, Midwife, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ayse Gul KOCA
Record Dates: First submitted 2023-07-08; First posted 2023-07-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Web-based Breastfeeding Counseling
Keywords: Breastfeeding counseling; Breastfeeding motivation; Web-based; Breast milk; Breastfeeding problems

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based breastfeeding counseling/experimental group (Experimental): The web-based breastfeeding counseling/experimental group (n =33) will be given the web-based breastfeeding counseling.
  Interventions: Other: The web-based breastfeeding counseling
- Control group (No Intervention): It will only take routine treatment and midwifery care.

INTERVENTIONS:
Other: The web-based breastfeeding counseling — To the web-based breastfeeding counseling/experimental group (n =33), during the first 6 months after birth, they will be directed to the web-based breastfeeding consultancy website. On this page, mothers will receive counseling on breastfeeding (written, visual, audio materials and telephone counseling) from birth. In addition, the Web-based breastfeeding counseling/experimental group will fill out data collection forms in the first 24 hours, 1st, 2nd, 4th and 6th months after delivery.
  Arms: Web-based breastfeeding counseling/experimental group

SUMMARY:
This randomized controlled study evaluates the effect of Web-Based Breastfeeding Counseling given to mothers on breastfeeding exclusively with breast milk in the first 6 months, breastfeeding motivation and breastfeeding problems.The main hypotheses it aims to answer are:

1. The web-based breastfeeding counseling given to the mothers in the experimental group is effective on the breastfeeding only for the first six months.
2. The web-based breastfeeding counseling given to the mothers in the experimental group is effective on the breastfeeding motivation of the mothers.
3. The web-based breastfeeding counseling given to the mothers in the experimental group is effective on the breastfeeding problems of the mothers.

DETAILED DESCRIPTION:
In the study, 66 mother will randomly assigned to web-based breastfeeding counseling/experimental group and control group. To the web-based breastfeeding counseling/experimental group (n =33), during the first 6 months after birth, they will be directed to the web-based breastfeeding consultancy website. On this page, mothers will receive counseling on breastfeeding (written, visual, audio materials and telephone counseling) from birth. On the other hand, no other intervention will be applied to the control group other than routine treatment and midwifery care. The primary outcome of the research is the effect of web-based breastfeeding counseling on the breastfeeding only for the first six months of mothers. The secondary outcome of the study is to determine the effect of web-based breastfeeding counseling on the breastfeeding motivation of the mothers. The tertiary outcome of the study is to determine the effect of web-based breastfeeding counseling on the breastfeeding problems of the mothers.

ELIGIBILITY:
Inclusion Criteria:

* treated at the relevant hospital
* who volunteered to participate in the research
* in the age range of 18-40
* oriented to place, time and person
* 37-42 weeks of pregnancy. between the weeks
* having first pregnancy
* having a healthy pregnancy
* Those who do not have any health problems that prevent breastfeeding (HIV, drug use, etc.)
* who is literate
* able to use computer or smart phone
* Those who do not have a communication barrier (not knowing Turkish, mental retardation, etc.)
* with internet at home

Exclusion Criteria:

* any health problem that prevents breastfeeding
* having a baby with any health problem that prevents breastfeeding
* who have a baby who was taken to the intensive care unit due to postpartum health problems
* with multiple pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Web-based breastfeeding counseling will be given to mothers after birth.
Enrollment: 66 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Postpartum Breastfeeding Evaluation and Follow-up Form | Change from before implementation (within the first 24 hours postpartum) and 1st, 2nd, 4rd and 6th months postpartum
  In this form, which was created by the researchers to evaluate and monitor postpartum breastfeeding, using the literature, there are questions that evaluate situations such as "the way babies are fed, the status of giving additional nutrients other than breast milk, the mothers' breastfeeding problems, and the mother's desire to continue breastfeeding.

SECONDARY OUTCOMES:
Breastfeeding Motivation Scale | Change from before implementation (within the first 24 hours postpartum) and 1st, 2nd, 4rd and 6th months postpartum
  It was developed by Kestler, Peleg et al (2015) and adapted into Turkish by Mızrak and Özerdoğan (2017). The scale consists of 24 items in total and consists of 5 sub-dimensions: "Integrated regulation" "intrinsic motivation and identified regulation", "introjected regulation - social approval", "introjected regulation - social pressure", and "external regulation - additional benefits".The Cronbach alpha value of the scale was found to be 0.855. Cronbach's alpha values for sub-dimensions vary between (0.846 - 0.670). The scale is in 4-point Likert type, and each item is scored between 1-4 (from 1 = "I strongly disagree" to 4 = "I totally agree"). The scale does not have a total score. The scores of the sub-dimensions are calculated by taking the average of the sub-dimension scores of the scale. As the score obtained from the scale sub-dimension increases, the motivation to breastfeed, which represents that sub-dimension, also increases.
Breastfeeding Problems Assesment Scale | Change from before implementation (within the first 24 hours postpartum) and 1st, 2nd, 4rd and 6th months postpartum
  It was developed by Wambach (1990), is a 30-item scale in order to determine the level of the problem experienced ("never happened" (1) to "unbearably happened" (5)). The total score of the scale varies between 18 and 90. A high score indicates that the severity of the problem has increased. The 18 items in the scale include mechanical concerns, process concerns, concerns about milk insufficiency , concerns about the udder and questions related to social concerns. The last 12 items of the scale evaluate whether breastfeeding is continued, whether formula is added, how often formula is given, and what are the breastfeeding difficulties related to the mother's decision to wean in case of early weaning. The Turkish validity and reliability of the scale was performed by Uyanık (2019) and he Cronbach's alpha value of the scale was found to be 0.77 for the sub-dimensions, and between 0.71-0.85.

CONTACTS AND LOCATIONS:
Overall Officials: Mine YURDAKUL, Doctorate, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)